CLINICAL TRIAL: NCT04288479
Title: Acute Effects of HIT on Fetal Well-being and Blood Flow Distribution - a Pilot Study
Brief Title: Acute Effects of High Intensity Training in Pregnancy on Fetal Well-being and Blood Flow Distribution
Acronym: HITFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62993
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy
Keywords: Exercise; High Intensity Interval Training; Pregnancy Outcome; Placental Circulation; Fetal Blood; Heart Rate, Fetal
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: before-after intervention effect measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doing a single HIT session in gestational week 22-36 (Experimental)
  Interventions: Behavioral: Single high-intensity interval training session

INTERVENTIONS:
Behavioral: Single high-intensity interval training session — 10 minutes warming up at low-to-moderate intensity, 8x30 seconds high intensity interval training with fetal heart rate measurement after each 30 second work-bout, 2 minutes recovery at low-to-moderate intensity. Continuous monitoring of maternal heart rate.
  Other Names: HIT

SUMMARY:
Pregnant women are recommended to be physically active ≥150 min/week, but <15% of Norwegian women attain this goal. Several well-designed studies on lifestyle interventions focusing primarily on exercise training in overweight/obese pregnant women have reported disappointing outcomes with regard to maternal glycemic control, gestational weight gain and infant outcomes. Low adherence to the training program was found to be a problem; the participants did not enjoy the exercise program and had difficulties scheduling time to exercise. Pregnant women also report that they are not sure what exercises are safe during pregnancy.

High intensity interval training (HIT), defined as short periods of intense activity separated by low-intensity breaks, has proved to induce superior improvements in insulin sensitivity and fitness compared with continuous moderate intensity training in individuals at increased risk for cardiometabolic diseases. Even short-term (6 weeks) HIT with brief (15-60 sec) work-bouts and a total time commitment of <45 min per week, improves insulin sensitivity similar to that attained after 6 months of traditional endurance training.

HIT is feasible and enjoyable for individuals with low fitness level and with obesity.

HIT is therefore a highly potent intervention that elicits important changes in a range of clinically relevant health outcomes in reproductive-aged women.

This study will investigate fetal responses to a single bout of HIT. Preliminary data of the investigators suggest that HIT does not negatively influence fetal heart rate. Others have reported that uterine and umbilical blood flow are not changed during or following acute exercise. However, no previous study has determined the acute effect of HIT on uterine blood flow and there are no studies investigating the fetal blood flow distribution in response to exercise. Since the relative distribution of blood to the fetal liver is associated with newborn adiposity, fetal blood flow distribution in response to exercise can provide insight about the effect of maternal exercise on offspring health.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, gestational week 22-36
* singleton fetus
* no known diseases
* capable of cycling on an ergometer bike

Exclusion Criteria:

* hypertension
* gestational diabetes mellitus
* any contraindication to exercise training

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
blood flow in fetal veins | 1 day
  examined by Doppler ultrasound during 30 minutes
blood flow in fetal arteries | 1 day
  examined by Doppler ultrasound during 30 minutes

SECONDARY OUTCOMES:
maternal heart rate | 1 dag
Fetal heart rate | 1 day
Umbilical vein diameter | 1 day
Maternal systolic blood pressure | 1 day
Maternal diastolic blood pressure | 1 day
Maternal body weight | 1 day
Maternal height | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Å Salvesen, md prof, Study Director — St Olavs Hospital, Dept of Obstetrics and Gynecology; Trine Moholdt, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Dept Circulation and Medical Imaging, EXCAR Exercise Lab, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No